CLINICAL TRIAL: NCT07034573
Title: Evaluation of the Performance of the Ventilation-filtration System for Operating Rooms at the Protestant Hospital of Mbouo-Bandjoun (VENTI-MBOUO)
Brief Title: Evaluation of a Ventilation-filtration System for Operating Rooms at the Protestant Hospital of Mbouo (VENTI-MBOUO)
Acronym: VENTI-MBOUO
Status: Completed | Type: Observational
Sponsor: Christian Doll (Other)
Collaborators: Universite Evangelique du Cameroun (Other); Paix et Santé - Gesundheit und Frieden global e.V. (Unknown)
Responsible Party: Sponsor-Investigator, Christian Doll, Dr., Universite Evangelique du Cameroun
Organization: Universite Evangelique du Cameroun (Other)
Other Study IDs: VENTI-MBOUO
Record Dates: First submitted 2025-06-02; First posted 2025-06-24 (Actual); Last update posted 2025-06-24 (Actual); Status verified 2025-06

CONDITIONS: Surgical Site Infections; Infections
Keywords: operating theatre; mechanical ventilation; air filtration; low resource context
MeSH Terms: conditions — Surgical Wound Infection; Infections | interventions — Operating Rooms

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- No patients, only a technical/microbial assessment of the ventilation-filtration system: No patients, only a technical/microbial assessment of the ventilation-filtration system in the operating theatre, with no contact with patients; therefore no "participant group/cohort"
  Interventions: Other: context adapted air filtration system for operating theatre

INTERVENTIONS:
Other: context adapted air filtration system for operating theatre — This observational pilot study combines a retrospective design (technical data) and a prospective design (microbial data) to evaluate a new air filtration system adapted to the context. For this research, the technical data of the system concerning air velocity, temperature, etc. will be used retrospectively. Microbial sampling in the operating theatre will be carried out prospectively.
  No patient contact will take place.

SUMMARY:
This research project is evaluating an air filtration system that is supposed to be adapted to the context, highly efficient and affordable. This air filtration system for operating theatres has been in use at Mbouo-Bandjoun hospital in Cameroon since 2019, with no incidents recorded to date.

In this proposed research project, only the ventilation system will be tested technically and microbiologically; no research will be carried out directly on patients or with patient participation.

Therefore, the research project is not expected to have any impact on patients. Technical test data will be evaluated retrospectively, while microbiological data will be collected prospectively without patient contact.

The air filtration system was installed in the OT of the Protestant hospital Mbouo (Hôpital Protestant de Mbouo) in 2019. Before the installation of the air filtrations system, the OT used window-based ventilation which seems, besides wall-mounted air conditioning systems, quite common in OT in Cameroonian hospitals.

The air filtrations system has been in regular use for 3.5 years before the first maintenance could be performed, due to COVID travel restrictions. This maintenance and technical measurement took place in November 2023.

Microbial samples in the OT were collected in Mai 2024. The data of the maintenance and technical measurements of the air filtration system are retrospectively used for this study. The parameters that are extracted from the maintenance documents are: particle counts, temperature, humidity, air velocity and pressure differences at various measurement points inside and outside the OT as well as inside the air filtration device.

To study the microbial burden in the OT, a prospective evaluation was carried out: In a time slot when no surgical procedures were planned, a passive sampling with settling plates was carried out.

DETAILED DESCRIPTION:
Abstract

The research project is entitled "Evaluation of the performance of the ventilation-filtration system for operating rooms at the Protestant Hospital of Mbouo-Bandjoun (VENTI-MBOUO)".

This research project evaluates an air filtration system supposedly adapted to the context, assumed to be very effective and at low cost. This operating theater air filtration system has been used at Mbouo-Bandjoun hospital for almost 4 years, without any incident problems having been recorded so far.

In this proposed research project, only the filtration-ventilation system will be tested technically and microbiologically; no research will be carried out directly on patients or with patient participation.

Therefore, the research project is not expected to have any impact on patients. Technical test data will be evaluated retrospectively, microbiological data will be collected prospectively in May 2024, without contact with the patient.

Introduction: Clean air in the operating theatre (OT) is crucial for safe surgery, to prevent surgical site infections. Air filtration devices are standard in most OT as required by international guidelines and regulations. However in low-ressource settings, common air filtration devices are only scarcely found in OT, mainly due to high cost; context-adapted low-cost solutions are urgently needed but not available.

Methods: A low-cost, supposedly high-efficient air filtration device was developed, adapted to the low-resource setting of a district hospital in Cameroon (l'Hôpital Protestant de Mbouo), constructed locally and implemented in 2019. An evaluation was done after nearly 4 years of regular use.

Variables to be evaluated:

Retrospectivey: The particle count in the operating room. Necessary maintenance in the last 3 years. Air velocity, air pressure, air direction in the operating room and in the air filtration device.

Prospectively: Changes in microbial air contamination in the operating room after turning on the device (during idle time, without any patient contact)

1. Introduction Surgical site infections (SSIs) are a significant health problem in low- and middle-income countries, leading to increased costs, prolonged hospital stays and disabilities. Up to one-third of patients undergoing surgery in Africa may be affected by SSI.

   One of the measures for preventing SSI is mechanical air filtration in operating theatres (OTs), which is the most commonly used method for purifying air in OTs in high-income countries. The two main mechanical filtration systems are turbulent mixed airflow ventilation and laminar airflow ventilation. These 'standard' systems in OT in high-income countries are expensive, often exceeding €50,000 in installation costs. This high cost may be an important reason why mechanical air filtration systems are not a common standard in low- and middle-income countries. Due to budget constraints, hospitals with limited resources may prefer simple air conditioning systems that are not suitable for use in OT or simply window ventilation, resulting in high bacterial loads in OT air.

   Context-appropriate solutions for clean air in OT in low-resource settings are therefore urgently needed. To our knowledge, this pilot study is the first in the world to evaluate a low-cost mechanical air filtration system that is believed to be highly effective and context-appropriate for OT in low-resource settings. This operating theatre air filtration system has been in use at the Mbouo-Bandjoun Hospital for almost four years, with no incidents reported to date.

   In this proposed research project, only the ventilation-filtration system will be tested technically and microbiologically; no research will be conducted directly on patients or with patient participation.

   Therefore, the research project should not have any impact on patients. Technical test data will be evaluated retrospectively, and microbiological data will be collected prospectively in May 2024, without contact with patients.
2. Research question (if applicable) What are the technical characteristics of the air ventilation-filtration system in the operating theatre of the Protestant Hospital in Mbouo? How effective is the ventilation-filtration system in reducing physical particles and microbiological contamination?
3. Research hypothesis(es) (if applicable)
4. Study objectives 4.1. General objective To evaluate the ventilation-filtration system in the operating theatre at the Protestant Hospital in Mbouo 4.2. Specific objectives

1. To evaluate the technical details of this system, including its particle filtration efficiency 2. To evaluate the reduction in microbes in the operating theatre achieved by this system 3. To compare the performance of this system with international standards

ELIGIBILITY:
Inclusion Criteria:

* No patients, only a technical/microbial assessment of the ventilation-filtration system in the operating theatre, with no contact with patients; therefore no source population and no inclusion criteria

Exclusion Criteria:

* No patients, only a technical/microbial assessment of the ventilation-filtration system in the operating theatre, with no contact with patients; therefore no source population and no exclusion criteria

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: No patients, only a technical/microbial assessment of the ventilation-filtration system in the operating theatre, with no contact with patients; therefore no study population
Sampling Method: Non-Probability Sample
Enrollment: 1 (Actual)
Dates: Start 2024-05-29 (Actual); Primary Completion 2024-05-31 (Actual); Study Completion 2024-05-31 (Actual)

PRIMARY OUTCOMES:
number of particles in the operating room air | retrospective: 4 years before study start
  The number of particles in the operating room air (particles per litre of air). Retrospective variable.
maintenance frequency | retrospective: 4 years before study start
  Maintenance of the ventilation-filtration system carried out over the last 4 years (frequency). Retrospective variable
system breakdowns | retrospective: 4 years before study start
  Number of system breakdowns. Retrospective variable
air speed and direction | retrospective: 4 years before study start
  Air speed (m/s) and air direction in the operating theatre and in the air filtration system.Retrospective variable
air pressure | retrospective: 4 years before study start
  air pressure (kPa) in the operating theatre and in the air filtration system.Retrospective variable
microbial air contamination | prospective: 29 april to 31 april 2024
  Changes in microbial contamination of the air in the operating theatre after the ventilation-air filtration system was switched on, during periods of inactivity in the operating theatre, without any contact with the patient (colony-forming units per Petri dish).Prospective variable

CONTACTS AND LOCATIONS:
Overall Officials: Christian Doll, Dr., Principal Investigator — Hessing Stiftung Orthopädische Fachkliniken
Locations (1):
- Mbouo Protestant Hospital, Bafoussam, Cameroon

IPD SHARING:
Plan to Share IPD: Yes
IPD that underlie the results reported (after deidentification) will be available beginning immediately after the article publication and ending 24 months after article publication. The data will be shared to researchers that provide a methodologically sound proposal, to achieve aims in the approved proposal. Corresponding author should be contacted.
Supporting Information: Study Protocol, SAP
Time Frame: for 24 months after article publication
Access Criteria: The data will be shared to researchers that provide a methodologically sound proposal, to achieve aims in the approved proposal. Corresponding author should be contacted.

REFERENCES:
- [Background] Hirsch T, Hubert H, Fischer S, Lahmer A, Lehnhardt M, Steinau HU, Steinstraesser L, Seipp HM. Bacterial burden in the operating room: impact of airflow systems. Am J Infect Control. 2012 Sep;40(7):e228-32. doi: 10.1016/j.ajic.2012.01.007. Epub 2012 Apr 26. PMID 22542026
- [Background] Pereira M, Tribess A, Buonanno G, Stabile L, Scungio M, Baffo I. Particle and Carbon Dioxide Concentration Levels in a Surgical Room Conditioned with a Window/Wall Air-conditioning System. Int J Environ Res Public Health. 2020 Feb 13;17(4):1180. doi: 10.3390/ijerph17041180. PMID 32069790
- [Background] Zhang B, Li L, Yao X, Gong Y, Zhang Y, Yang H, Li W, Lin L, Yang Y, Zhang H, Jia H. Analysis of Air Purification Methods in Operating Rooms of Chinese Hospitals. Biomed Res Int. 2020 Feb 1;2020:8278943. doi: 10.1155/2020/8278943. eCollection 2020. PMID 32076617